CLINICAL TRIAL: NCT01268488
Title: Clinical Trial Protocol for NINJA 2 System With CONTOUR Sensor
Brief Title: Performance of an Investigational Blood Glucose Monitoring System in a Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2010-008-02
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Results first posted 2012-10-16 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the System (Experimental): Untrained subjects with diabetes obtained capillary fingerstick, palm, and forearm blood and performed Blood Glucose (BG) tests using a Ninja 2 investigational blood glucose meter and the Contour® sensor. This BG monitoring system will not proceed to marketed product.
  Interventions: Device: Ninja 2 Investigational Blood Glucose Meter

INTERVENTIONS:
Device: Ninja 2 Investigational Blood Glucose Meter — Untrained subjects with diabetes performed Blood Glucose(BG) tests from the subject's capillary blood obtained from fingerstick, palm, and forearm using the Ninja 2 investigational meter. All BG results were compared to a reference laboratory glucose method. Subjects' success at performing basic tasks using only the User Guide were rated by study staff.

SUMMARY:
The purpose of this study is to evaluate the performance of an investigational blood glucose meter with the Contour sensor strip. It was decided that this investigational monitoring system would not be part of a regulatory submission and it will not proceed to marketed product.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and above
* Type 1 or type 2 diabetes
* Currently self-testing blood glucose at home at least twice daily
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Currently Pregnant
* Hemophilia or any other bleeding disorder
* Employee of competitive medical device company
* Cognitive disorder or other condition which, in the opinion of the investigator, would put the person at risk or seriously compromise the integrity of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Caswell, PhD, Principal Investigator — Consumer Product Testing Company
Locations (1):
- Consumer Product Testing Company, Fairfield, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended Users of the System: Untrained subjects with diabetes obtained capillary fingerstick, palm, and forearm blood and performed Blood Glucose (BG) tests using a Ninja 2 investigational blood glucose meter and the Contour® sensor.
  Ninja 2 Investigational Blood Glucose Meter : Untrained subjects with diabetes performed Blood Glucose(BG) tests from the subject's capillary blood obtained from fingerstick, palm, and forearm using the Ninja 2 investigational meter. All BG results were compared to a reference laboratory glucose method. Subjects' success at performing basic tasks using only the User Guide were rated by study staff.
Period: Overall Study
Arm/Group | Intended Users of the System
Started | 98
Completed | 93
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 98
Age, Continuous [Mean (Full Range); unit: years] | 50.8 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 45
Region of Enrollment [Number; unit: participants]
  United States | 98

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Fingerstick Blood Glucose (BG) Results Within +/- 5 to 15mg/dL (<75 mg/dL) or Within +/- 5% to 20% (>=75 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes tested subject fingerstick blood using an investigational blood glucose meter (BGM). BGM results were compared to a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG results were used to calculate the number of BG results within +/- 5 to 15 mg/dL (for reference BG results <75mg/dL) or +/- 5 to 20% (for reference BG results >=75mg/dL) of the reference method results.
Time Frame: 2 hours
Population: 178 BG results possible-88 subjects tested 2 strip lots(88x2)/2 subjects had 1 reading(2x1). Withdrawn by Principal Investigator(PI)-3 subjects experienced Adverse Events before performance testing / one subject did not meet inclusion/exclusion. Data from 4 subjects were not evaluable since exceeded time between meter testing and reference method.
Measure: Number; unit: Number of BG Test Results
Units Other Than Participants: BG test results
Groups:
- Intended Users of the System: Untrained subjects with diabetes obtained capillary fingerstick, palm, and forearm blood and performed Blood Glucose (BG) tests using a Ninja 2 investigational blood glucose meter and the Contour® sensor.
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 90
Number analyzed (BG test results) | 178
Number of BG Test Results
  # within +/-15mg/dL (<75mg/dL) or 20% (>=75mg/dL) | 172
  # within +/-15mg/dL (<75mg/dL) or 15% (>=75mg/dL) | 171
  # within +/-10mg/dL (<75mg/dL) or 10% (>=75mg/dL) | 155
  # within +/-5mg/dL (<75mg/dL) or 5% (>=75mg/dL) | 88

2. Secondary Outcome: Numbers of Palm Blood Glucose (BG) Results Within +/- 5 to 15 mg/dL (<75 mg/dL) or Within +/- 5% to 20% (>=75 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes used an investigational blood glucose meter (BGM) with subject capillary blood obtained from the palm. BGM results were compared to a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG results were used to calculate the number of BG results within +/- 5 to 15 mg/dL (for reference BG results <75mg/dL) or +/- 5% to 20% (for reference BG results >=75mg/dL) of the reference method results.
Time Frame: 2 hours
Population: 161 BG results-80 subjects tested 2 strip lots;1 subject had 1 reading. Withdrawn by PI- 3 subject Adverse Events before performance testing;1 subject did not meet inclusion/exclusion. 6 subjects- Data not evaluable:exceeded time between meter testing and reference method. 7 subjects-Low bg results disallowed palm testing per protocol.
Measure: Number; unit: Number of BG Test Results
Units Other Than Participants: Number of BG test results
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 81
Number analyzed (Number of BG test results) | 161
Number of BG Test Results
  # within +/-15mg/dL (<75mg/dL) or 20% (>=75mg/dL) | 150
  # within +/-15mg/dL (<75mg/dL) or 15% (>=75mg/dL) | 136
  # within +/-10mg/dL (<75mg/dL) or 10% (>=75mg/dL) | 97
  # within +/-5mg/dL (<75mg/dL) or 5% (>=75mg/dL) | 57

3. Secondary Outcome: Number of Subjects Rated as<=3 Performing Basic Meter Tasks (Labeling Comprehension)
Description: Subjects reviewed the instructions for use (User Guide and Quick Reference Guide) to learn to use the system. Study staff then observed and rated the subjects(1 to 4) on their success at performing the tasks. Scale: 1.Success in performing tasks correctly without assistance. 2.Successful with additional review of User Guide. 3.Successful with additional review and study staff assist similar to review of a specific function during a Customer Service call. 4.Subject did not perform task correctly and study staff intervention was required.
Time Frame: 2 hours
Population: 97 participants analyzed: one subject was found not to meet inclusion/exclusion criteria so subject was withdrawn and no data from this subject was evaluated. For palm and forearm testing tasks, 2 additional subjects (with nonevaluable BG data) were not included. Only 95 participants were rated for those particular tasks.
Measure: Number; unit: participants
Groups:
- Intended Users of the System: Ninja 2 Investigational Blood Glucose Meter : Untrained subjects with diabetes performed Blood Glucose(BG) tests from the subject's capillary blood obtained from fingerstick, palm, and forearm using the Ninja 2 investigational meter. All BG results were compared to a reference laboratory glucose method. Subjects' success at performing basic tasks using only the User Guide were rated by study staff.
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 97
participants
  Turn meter on / off | 96
  Date and time set on meter | 87
  Normal control testing | 93
  Subject blood testing - fingerstick | 91
  Subject blood testing - palm (of 95) | 85
  Subject blood testing - forearm (of 95) | 65

4. Secondary Outcome: Numbers of Forearm Blood Glucose (BG) Results Within +/- 5 to 15 mg/dL (<75 mg/dL) or Within +/- 5% to 20% (>=75 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes used an investigational blood glucose meter (BGM) with subject capillary blood obtained from the forearm. BGM results were compared to a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG results were used to calculate the number of BG results within +/- 5 to 15 mg/dL (for reference BG results <75mg/dL) or +/- 5% to 20% (for reference BG results >=75mg/dL) of the reference method results.
Time Frame: 2 hours
Population: 158 BG results-78 subjects tested 2 strip lots;2 subjects tested 1 strip lot. 7 subjects-Low BG results disallowed forearm testing per protocol. 1 subject-Missing data. Remainder same as 'palm' analysis population description.
Measure: Number; unit: Number of BG Test Results
Units Other Than Participants: Number of BG Test Results
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 80
Number analyzed (Number of BG Test Results) | 158
Number of BG Test Results
  # within +/-15mg/dL (<75mg/dL) or 20% (>=75mg/dL) | 147
  # within +/-15mg/dL (<75mg/dL) or 15% (>=75mg/dL) | 133
  # within +/-10mg/dL (<75mg/dL) or 10% (>=75mg/dL) | 99
  # within +/-5mg/dL (<75mg/dL) or 5% (>=75mg/dL) | 56

ADVERSE EVENTS:
Arm/Group | Intended Users of the System
Serious Adverse Events (participants affected / at risk) | 0/98
Other Adverse Events (participants affected / at risk) | 0/98

LIMITATIONS AND CAVEATS:
It was decided that this investigational BG monitoring system would not be part of a regulatory submission. It will not proceed to market.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days